CLINICAL TRIAL: NCT00977964
Title: Tolerance of Healthy Term Infants Fed Infant Formulas
Brief Title: Tolerance of Healthy Term Infants Fed Infant Formulas #3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie L Swearengin, RN, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK70
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Gastrointestinal Tolerance
Keywords: Infant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Milk Based Protein Formula Process A (Experimental)
  Interventions: Other: Experimental milk protein infant formula Process A
- Milk Based Protein Formula Process B (Experimental)
  Interventions: Other: Experimental milk protein infant formula Process B
- Milk Based Protein Formula Process C (Experimental)
  Interventions: Other: Experimental milk protein infant formula Process C
- Milk Based Protein Formula Process D (Experimental)
  Interventions: Other: Experimental milk protein infant formula Process D
- Milk Based Protein Formula Process E (Experimental)
  Interventions: Other: Experimental milk protein infant formula Process E
- Milk Based Protein Formula Process F (Experimental)
  Interventions: Other: Experimental milk protein infant formula Process F

INTERVENTIONS:
Other: Experimental milk protein infant formula Process A — ad lib for 1-8 days of age until 28 days of age
  Arms: Milk Based Protein Formula Process A
Other: Experimental milk protein infant formula Process B — ad lib from 1-8 days of age until 28 days of age
  Arms: Milk Based Protein Formula Process B
Other: Experimental milk protein infant formula Process C — ad lib from 1-8 days of age to 28 days of age
  Arms: Milk Based Protein Formula Process C
Other: Experimental milk protein infant formula Process D — ad lib from 1-8 days of age until 28 days of age
  Arms: Milk Based Protein Formula Process D
Other: Experimental milk protein infant formula Process E — ad lib from 1-8 days of age until 28 days of age
  Arms: Milk Based Protein Formula Process E
Other: Experimental milk protein infant formula Process F — ad lib from 1-8 days of age until 28 days of age
  Arms: Milk Based Protein Formula Process F

SUMMARY:
The primary objective of this study is to assess the comparative gastrointestinal (GI) tolerance of normal term infants to six experimental milk protein-based powdered infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Infant is judged to be in good health.
* Infant is a singleton from a full term birth.
* Infant's birth weight was > 2490 g (~5 lbs 8 oz.
* Infant is between 0 and 8 days of age at enrollment.
* Infants using medications, home remedies ,herbal preparations or rehydration fluids that might affect GI tolerance may not be enrolled.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study, unless instructed otherwise by their healthcare professional.

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Infant has been treated with antibiotics.
* Infant has received probiotics.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary variable is Gastrointestinal tolerance. | 1-28 days of age

SECONDARY OUTCOMES:
The secondary variables are additional measures of GI tolerance and parental feedback. | 1-28 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Caude T Ashley, MD, Principal Investigator — Alabama Clinical Therapeutics, LLC; Terri L Ashmeade, MD, Principal Investigator — USF Department of Pediatrics; Jay Cohen, MD, Principal Investigator — Discovery Clinical Research, Inc.; Timothy Crum, MD, Principal Investigator — Rockwood Clinic; Cole Ezeoke, MD, Principal Investigator — North Georgia Clinical Research, White's Pediatrics; Sharon Groh-Wargo, PhD, RD, LD, Principal Investigator — MetroHealth Medical Center; James Guerrieri, MD, Principal Investigator — Institute of Clinical Research, LLC; James Hedrick, MD, Principal Investigator — Kentucky Pediatric Research; Jeffrey Hirschfield, MD, Principal Investigator — SCORE Physician Alliance, LLC; Kevin Mullen, MD, Principal Investigator — Medical Associates Clinic, PC; Chris Peltier, MD, Principal Investigator — Pediatric Associates of Mount Carmel, Inc.; Martin J Schear, MD, Principal Investigator — Dayton Clinical Research; Julie Shepard, MD, Principal Investigator — Ohio Pediatric Research Association; William Stepp, MD, Principal Investigator — Sarah Cannon Research Institute, LLC; L Louise Tetrick, MD, Principal Investigator — Northpoint Pediatrics
Locations (15):
- United States (15):
  - Alabama Clinical Therapeutics, Dothan, Alabama
  - All Women's Heatlthcare of West Broward, Inc: Discovery Clinical Research, Inc, Plantation, Florida
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - North Georgia Clinical Research, Dalton, Georgia
  - Northpoint Pediatrics, LLC, Indianapolis, Indiana
  - Medical Associates Clinic, PC, Dubuque, Iowa
  - Kentucky Pediatric / Adult Research, Bardstown, Kentucky
  - Pediatric Associates of Mount Carmel, Inc, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association, Inc., Huber Heights, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Rockwood Clinic North - Pediatrics, Spokane, Washington

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831